CLINICAL TRIAL: NCT03480763
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by Administration of PNEUMOVAX™23 One Year Later in Healthy Adults 50 Years of Age or Older (PNEU-PATH)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by PNEUMOVAX™23 in Healthy Adults 50 Years of Age or Older (V114-016/PNEU-PATH)
Acronym: PNEU-PATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-016; V114-016 (Other: Merck Protocol Number); 2017-004024-30 (EudraCT Number)
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2)
  Interventions: Biological: V114; Biological: PNEUMOVAX™23
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2)
  Interventions: Biological: Prevnar 13™; Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and Merck Aluminum Phosphate Adjuvant (125 mcg) in each 0.5 mL dose
  Arms: V114
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose
  Other Names: PCV13
  Arms: Prevnar 13™
Biological: PNEUMOVAX™23 — 23-valent pneumococcal polysaccharide vaccine with serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F (25 mcg each) in each 0.5 mL dose
  Other Names: PPV23

SUMMARY:
This study is designed 1) to evaluate the safety, tolerability, and immunogenicity of V114 and Prevnar 13™, 2) to describe the safety of sequential administration of V114 or Prevnar 13™ followed by PNEUMOVAX™23, and 3) to evaluate the immune responses to the 15 serotypes contained in V114 when PNEUMOVAX™23 is given approximately 12 months after receipt of either V114 or Prevnar 13™ in healthy adults 50 years of age or older. There was no formal hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good health
* Female participant: not pregnant, not breastfeeding and 1) not of childbearing potential, or 2) of childbearing potential and agrees to practice contraception through 6 weeks after administration of last study vaccine.

Exclusion Criteria

* History of invasive pneumococcal disease
* Known hypersensitivity to any component of pneumococcal polysaccharide vaccine, pneumococcal conjugate vaccine, or any diphtheria toxoid-containing vaccine.
* Known or suspected impairment of immune function
* Coagulation disorder contraindicating intramuscular vaccination
* History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Female participant: positive urine or serum pregnancy test
* Prior administration of any pneumococcal vaccine
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention at least 30 days before study entry.
* Received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination. (Note: Topical, ophthalmic, intra-articular or soft-tissue [e.g., bursa, tendon steroid injections], and inhaled/nebulized steroids are permitted).
* Received immunosuppressive therapy
* Received a blood transfusion or blood products within 6 months of enrollment
* Participated in another clinical study of an investigational product within 2 months of enrollment
* Current user of recreational or illicit drugs or history of drug or alcohol abuse or dependence.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- United States (15):
  - East Valley Family Physicians ( Site 0104), Chandler, Arizona
  - Central Phoenix Medical Clinic, LLC ( Site 0125), Phoenix, Arizona
  - Encompass Clinical Research ( Site 0118), Spring Valley, California
  - Diablo Clinical Research, Inc ( Site 0132), Walnut Creek, California
  - Clinical Research of South Florida ( Site 0126), Coral Gables, Florida
  - QPS Miami Research Associates ( Site 0116), South Miami, Florida
  - Heartland Research Associates, Llc ( Site 0115), Wichita, Kansas
  - Centennial Medical Group ( Site 0109), Elkridge, Maryland
  - Rapid Medical Research, Inc. ( Site 0119), Cleveland, Ohio
  - University of Texas Medical Branch at Galveston ( Site 0127), Galveston, Texas
  - Texas Center For Drug Development ( Site 0107), Houston, Texas
  - Diagnostics Research Group ( Site 0100), San Antonio, Texas
  - J Lewis Research Inc / Foothill Family Clinic ( Site 0123), Salt Lake City, Utah
  - J Lewis Research Inc/Jordan River Family Medicine ( Site 0114), South Jordan, Utah
  - Health Research of Hampton Roads, Inc. ( Site 0106), Newport News, Virginia
- South Korea (2):
  - Seoul National University Hospital ( Site 0400), Seoul
  - Korea University Guro Hospital ( Site 0401), Seoul
- Spain (3):
  - CAP Centelles ( Site 0303), Centelles, Barcelona
  - Instituto de Ciencias Medicas.ICM ( Site 0301), Alicante
  - Fundacion Oftalmologica del Mediterraneo ( Site 0300), Valencia
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 0502), Dawan
  - National Taiwan University Hospital ( Site 0500), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Song JY, Chang CJ, Andrews C, Diez-Domingo J, Oh MD, Dagan R, Hartzel J, Pedley A, Li J, Sterling T, Tamms G, Chiarappa JA, Lutkiewicz J, Musey L, Tu Y, Buchwald UK; V114-016 (PNEU-PATH) study group. Safety, tolerability, and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, followed by sequential PPSV23 vaccination in healthy adults aged >/=50 years: A randomized phase III trial (PNEU-PATH). Vaccine. 2021 Oct 15;39(43):6422-6436. doi: 10.1016/j.vaccine.2021.08.038. Epub 2021 Sep 4. PMID 34489128
- [Derived] Huang L, Yang X, Li H, Xie Z, Zhu T, You W, Wang Z, Tan J, Feng G, Sun Q, Wang B, Han X, Wang Y. Immune persistence of a single dose of 23-valent pneumococcal polysaccharide vaccine: A 6-year follow-up. Hum Vaccin Immunother. 2025 Dec;21(1):2517489. doi: 10.1080/21645515.2025.2517489. Epub 2025 Jun 19. PMID 40537903

RESULTS

PARTICIPANT FLOW:
Groups:
- V114: Participants were to receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
- Prevnar 13™: Participants were to receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 327 | 325
Vaccination 1 - (V114 or Prevnar 13™, Day 1) | 326 | 325
Vaccination 2 - (PNEUMOVAX™23, Month 12) | 298 | 302
Completed | 303 | 306
Not Completed | 24 | 19
Not completed — Withdrawal by Subject | 18 | 10
Not completed — Lost to Follow-up | 4 | 7
Not completed — non-study pneumococcal vaccine | 1 | 0
Not completed — oncological treatment | 0 | 2
Not completed — pain with vaccination | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 327 | 325 | 652
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.0) | 64.1 (8.4) | 64.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 181 | 371
  Male | 137 | 144 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 37 | 79
  Not Hispanic or Latino | 283 | 287 | 570
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 103 | 103 | 206
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 22 | 40
  White | 203 | 198 | 401
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events Following V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following vaccination with V114 or Prevnar 13™, the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain.
Time Frame: Up to 5 days after Vaccination 1
Population: The analysis population included all randomized participants who received the relevant study vaccination for the timepoint of interest. (In the Prevnar 13™ group, 324 were vaccinated with Prevnar 13™; 1 was incorrectly vaccinated with V114.)
Measure: Number; unit: Percentage of Participants
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and were to receive a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and were to receive a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 327 | 324
Percentage of Participants
  Injection site redness/erythema | 9.8 | 5.6
  Injection site tenderness/pain | 55.0 | 41.4
  Injection site swelling | 16.2 | 11.4
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Injection site redness/erythema; Test type: Other — Estimated differences, confidence intervals (CIs), and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p = 0.043, Miettinen & Nurminen; Difference in Percent = 4.2, 95% CI 2-sided [0.1 to 8.5]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Injection site tenderness/pain; Test type: Other — Estimated differences, CIs, and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p < 0.001, Miettinen & Nurminen; Difference in Percent = 13.7, 95% CI 2-sided [6.0 to 21.2]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Injection site swelling; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.077, Miettinen & Nurminen; Difference in Percent = 4.8, 95% CI 2-sided [-0.5 to 10.2]

2. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events Following PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following vaccination with PNEUMOVAX™23, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue.
Time Frame: Up to 5 days after Vaccination 2
Population: The analysis population included all randomized participants who received the relevant study vaccination for the timepoint of interest.
Measure: Number; unit: Percentage of Participants
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 298 | 302
Percentage of Participants
  Injection site redness/erythema | 17.4 | 16.9
  Injection site tenderness/pain | 62.1 | 58.6
  Injection site swelling | 28.2 | 26.2
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Injection site redness/erythema; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.855, Miettinen & Nurminen; Difference in Percent = 0.6, 95% CI 2-sided [-5.5 to 6.6]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Injection site tenderness/pain; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.385, Miettinen & Nurminen; Difference in Percent = 3.5, 95% CI [-4.4 to 11.3]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Injection site swelling; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.577, Miettinen & Nurminen; Difference in Percent = 2.0, 95% CI 2-sided [-5.1 to 9.2]

3. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following vaccination with V114 or Prevnar 13™, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue.
Time Frame: Up to 14 days after Vaccination 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 327 | 324
Percentage of Participants
  Joint pain/arthralgia | 6.4 | 5.2
  Tiredness/fatigue | 23.5 | 13.9
  Headache | 14.1 | 12.7
  Muscle pain/myalgia | 17.7 | 11.1
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Joint pain/arthralgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.523, Miettinen & Nurminen; Difference in Percent = 1.2, 95% CI 2-sided [-2.5 to 4.9]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Tiredness/fatigue; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.002, Miettinen & Nurminen; Difference in Percent = 9.7, 95% CI 2-sided [3.7 to 15.6]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Headache; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.597, Miettinen & Nurminen; Difference in Percent = 1.4, 95% CI 2-sided [-3.9 to 6.7]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Muscle pain/myalgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.016, Miettinen & Nurminen; Difference in Percent = 6.6, 95% CI 2-sided [1.2 to 12.1]

4. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following PNEUMOVAX™23
Description: as for outcome 2
Time Frame: Up to 14 days after Vaccination 2
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 298 | 302
Percentage of Participants
  Joint pain/arthralgia | 8.4 | 8.3
  Tiredness/fatigue | 25.8 | 21.9
  Headache | 12.1 | 12.6
  Muscle pain/myalgia | 21.5 | 16.6
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Joint pain/arthralgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.961, Miettinen & Nurminen; Difference in Percent = 0.1, 95% CI 2-sided [-4.4 to 4.7]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Tiredness/fatigue; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.252, Miettinen & Nurminen; Difference in Percent = 4.0, 95% CI 2-sided [-2.8 to 10.8]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Headache; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.852, Miettinen & Nurminen; Difference in Percent = -0.5, 95% CI 2-sided [-5.8 to 4.8]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Muscle pain/myalgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.125, Miettinen & Nurminen; Difference in Percent = 4.9, 95% CI 2-sided [-1.4 to 11.2]

5. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events Following V114 or Prevnar 13™
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine will be determined by the investigator. Following vaccination with V114 or Prevnar 13™, the percentage of participants with vaccine-related serious adverse events was assessed.
Time Frame: Up to 12 months after Vaccination 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 327 | 324
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Vaccine-related SAEs following V114 or Prevnar 13™; Test type: Other — [test comment as in outcome 1, analysis 2]; Difference in Percent = 0.0, 95% CI 2-sided [-1.2 to 1.2]

6. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events Following PNEUMOVAX™23
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine will be determined by the investigator. Following vaccination with PNEUMOVAX™23, the percentage of participants with vaccine-related serious adverse events was assessed.
Time Frame: Month 12 to Month 13 (Up to 44 days after Vaccination 2)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 298 | 302
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Vaccine-related SAEs following PNEUMOVAX™23; Test type: Other — [test comment as in outcome 1, analysis 2]; Difference in Percent = 0.0, 95% CI 2-sided [-1.3 to 1.3]

7. Primary Outcome: Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity at 30 Days Following PNEUMOVAX™23
Description: Serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) (estimated) and GMT ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated. OPA for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using a Multiplexed Opsonophagocytic Assay.
Time Frame: Month 13 (30 days after Vaccination 2)
Population: The analysis population consisted of all randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and had sufficient data to perform the analyses.
Measure: Number; unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 392.2 | 283.2
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 322
  Serotype 3 (Shared) | 282.6 | 262.8
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 1671.9 | 1580.4
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 705.5 | 583.9
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 3261.5 | 2806.8
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 3223.9 | 2872.0
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 322
  Serotype 7F (Shared) | 5125.6 | 4848.0
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 2059.5 | 1872.0
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 3370.9 | 2660.5
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 2379.6 | 2103.9
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 3657.1 | 3170.8
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 2229.7 | 2156.2
  Serotype 23F (Shared): number analyzed (Participants) | 320 | 323
  Serotype 23F (Shared) | 1894.2 | 1485.1
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 3124.4 | 1921.6
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 7881.6 | 8269.9
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — Geometric mean titer (GMT) ratio and 95% confidence interval (CI) are estimated from a constrained longitudinal data analysis (cLDA) model; GMT Ratio = 1.38, 95% CI 2-sided [1.10 to 1.74]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.08, 95% CI 2-sided [0.90 to 1.29]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.06, 95% CI 2-sided [0.85 to 1.32]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.21, 95% CI 2-sided [0.94 to 1.56]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.16, 95% CI 2-sided [0.95 to 1.43]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.12, 95% CI 2-sided [0.93 to 1.35]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.06, 95% CI 2-sided [0.90 to 1.25]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.10, 95% CI 2-sided [0.91 to 1.33]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.27, 95% CI 2-sided [1.05 to 1.53]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.13, 95% CI 2-sided [0.95 to 1.34]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.15, 95% CI 2-sided [0.96 to 1.38]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.03, 95% CI 2-sided [0.89 to 1.20]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.28, 95% CI 2-sided [1.01 to 1.61]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.63, 95% CI 2-sided [1.29 to 2.06]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.95, 95% CI 2-sided [0.77 to 1.17]

8. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Immunoglobulin G at 30 Days Following PNEUMOVAX™23
Description: Serotype-specific Immunoglobulin G (IgG) geometric mean concentrations (GMCs) (estimated) and GMC ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMC ratios); within-group CIs were not calculated. IgG for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using an electrochemiluminescence assay.
Time Frame: Month 13 (30 days after Vaccination 2)
Population: as for outcome 7
Measure: Number; unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 5.21 | 5.68
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 3 (Shared) | 1.05 | 1.05
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 1.99 | 2.29
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 5.77 | 5.82
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 4.97 | 4.28
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 6.71 | 5.77
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 7F (Shared) | 5.99 | 6.06
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 4.96 | 4.75
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 14.82 | 12.72
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 7.31 | 6.29
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 13.10 | 11.88
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 9.38 | 8.62
  Serotype 23F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 23F (Shared) | 4.83 | 4.24
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 4.85 | 3.39
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 10.60 | 13.30
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — Geometric mean concentration (GMC) ratio and 95% confidence interval (CI) are estimated from a constrained longitudinal data analysis (cLDA) model; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.07]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.00, 95% CI 2-sided [0.87 to 1.16]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.87, 95% CI 2-sided [0.74 to 1.02]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.99, 95% CI 2-sided [0.84 to 1.18]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.16, 95% CI 2-sided [0.96 to 1.41]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.16, 95% CI 2-sided [0.96 to 1.40]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.99, 95% CI 2-sided [0.85 to 1.16]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.04, 95% CI 2-sided [0.89 to 1.22]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.17, 95% CI 2-sided [0.98 to 1.39]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.16, 95% CI 2-sided [1.00 to 1.36]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.10, 95% CI 2-sided [0.95 to 1.29]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.09, 95% CI 2-sided [0.93 to 1.27]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.14, 95% CI 2-sided [0.96 to 1.35]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.43, 95% CI 2-sided [1.16 to 1.77]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.80, 95% CI 2-sided [0.67 to 0.95]

9. Secondary Outcome: GMT of Serotype-specific OPA at Day 30
Description: Serotype-specific OPA GMTs (estimated) and GMT ratios with 95% CIs were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated. OPA for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using a Multiplexed Opsonophagocytic Assay.
Time Frame: Day 30
Population: as for outcome 7
Measure: Number; unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 361.6 | 296.2
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 322
  Serotype 3 (Shared) | 245.4 | 129.4
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 1280.4 | 1685.9
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 699.0 | 655.9
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 7352.8 | 6184.2
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 5958.1 | 3631.2
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 322
  Serotype 7F (Shared) | 4966.9 | 5207.6
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 2329.9 | 2293.0
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 2677.3 | 2458.1
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 4298.2 | 2896.3
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 4856.1 | 3783.0
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 2418.8 | 2203.5
  Serotype 23F (Shared): number analyzed (Participants) | 320 | 323
  Serotype 23F (Shared) | 2648.7 | 1726.9
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 3471.1 | 99.6
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 11392.4 | 1244.7
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.22, 95% CI 2-sided [0.94 to 1.58]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.90, 95% CI 2-sided [1.56 to 2.30]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.76, 95% CI 2-sided [0.60 to 0.97]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.07, 95% CI 2-sided [0.81 to 1.40]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.19, 95% CI 2-sided [0.92 to 1.53]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.64, 95% CI 2-sided [1.31 to 2.06]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.95, 95% CI 2-sided [0.80 to 1.14]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.02, 95% CI 2-sided [0.83 to 1.24]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.09, 95% CI 2-sided [0.87 to 1.37]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.48, 95% CI 2-sided [1.20 to 1.84]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.28, 95% CI 2-sided [1.06 to 1.55]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.10, 95% CI 2-sided [0.92 to 1.32]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.53, 95% CI 2-sided [1.18 to 2.00]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 34.86, 95% CI 2-sided [26.13 to 46.50]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 9.15, 95% CI 2-sided [7.48 to 11.20]

10. Secondary Outcome: GMC of Serotype-specific IgG at Day 30
Description: Serotype-specific IgG GMC (estimated) and GMC ratios with 95% CIs were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMC ratios); within-group CIs were not calculated. IgG for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using an electrochemiluminescence assay.
Time Frame: Day 30
Population: as for outcome 7
Measure: Number; unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 6.97 | 7.86
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 3 (Shared) | 1.02 | 0.59
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 2.36 | 2.98
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 5.43 | 5.21
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 11.48 | 8.22
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 13.69 | 8.35
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 7F (Shared) | 7.14 | 7.82
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 6.10 | 5.39
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 12.68 | 11.59
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 16.67 | 10.66
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 18.59 | 16.48
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 12.00 | 10.53
  Serotype 23F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 23F (Shared) | 9.76 | 6.07
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 5.07 | 0.31
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 14.31 | 1.12
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.89, 95% CI 2-sided [0.72 to 1.09]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.74, 95% CI 2-sided [1.46 to 2.07]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.79, 95% CI 2-sided [0.64 to 0.99]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.04, 95% CI 2-sided [0.84 to 1.30]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMCs, GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.40, 95% CI 2-sided [1.10 to 1.77]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.64, 95% CI 2-sided [1.28 to 2.10]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.91, 95% CI 2-sided [0.74 to 1.13]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.13, 95% CI 2-sided [0.91 to 1.41]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.09, 95% CI 2-sided [0.87 to 1.38]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.56, 95% CI 2-sided [1.27 to 1.92]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.13, 95% CI 2-sided [0.91 to 1.39]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.14, 95% CI 2-sided [0.92 to 1.41]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.61, 95% CI 2-sided [1.27 to 2.04]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 16.54, 95% CI 2-sided [13.78 to 19.86]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 12.82, 95% CI 2-sided [10.82 to 15.19]

11. Secondary Outcome: Geometric Mean Fold Rise in Serotype-specific OPA Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a Multiplexed Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 307 | 314
  Serotype 1 (Shared) | 22.3 [18.5 to 26.9] | 16.7 [13.8 to 20.2]
  Serotype 3 (Shared): number analyzed (Participants) | 305 | 313
  Serotype 3 (Shared) | 8.0 [6.9 to 9.2] | 4.4 [3.8 to 5.1]
  Serotype 4 (Shared): number analyzed (Participants) | 305 | 312
  Serotype 4 (Shared) | 18.3 [15.0 to 22.4] | 23.3 [19.3 to 28.3]
  Serotype 5 (Shared): number analyzed (Participants) | 310 | 315
  Serotype 5 (Shared) | 17.2 [14.2 to 20.9] | 16.2 [13.3 to 19.7]
  Serotype 6A (Shared): number analyzed (Participants) | 279 | 283
  Serotype 6A (Shared) | 17.4 [14.2 to 21.2] | 13.9 [11.5 to 16.8]
  Serotype 6B (Shared): number analyzed (Participants) | 302 | 306
  Serotype 6B (Shared) | 28.5 [23.1 to 35.2] | 18.4 [14.9 to 22.7]
  Serotype 7F (Shared): number analyzed (Participants) | 296 | 296
  Serotype 7F (Shared) | 10.7 [8.7 to 13.0] | 10.5 [8.5 to 13.1]
  Serotype 9V (Shared): number analyzed (Participants) | 299 | 310
  Serotype 9V (Shared) | 6.1 [5.2 to 7.1] | 5.6 [4.7 to 6.5]
  Serotype 14 (Shared): number analyzed (Participants) | 304 | 308
  Serotype 14 (Shared) | 6.6 [5.4 to 8.0] | 6.0 [4.9 to 7.4]
  Serotype 18C (Shared): number analyzed (Participants) | 301 | 310
  Serotype 18C (Shared) | 18.1 [15.1 to 21.7] | 12.2 [10.2 to 14.5]
  Serotype 19A (Shared): number analyzed (Participants) | 301 | 309
  Serotype 19A (Shared) | 13.4 [11.1 to 16.3] | 10.0 [8.4 to 12.0]
  Serotype 19F (Shared): number analyzed (Participants) | 298 | 308
  Serotype 19F (Shared) | 7.8 [6.7 to 9.2] | 6.4 [5.5 to 7.5]
  Serotype 23F (Shared): number analyzed (Participants) | 284 | 288
  Serotype 23F (Shared) | 18.8 [15.2 to 23.1] | 12.2 [9.8 to 15.2]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 250 | 249
  Serotype 22F (Unique to V114) | 32.5 [24.2 to 43.6] | 1.1 [0.8 to 1.4]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 305 | 298
  Serotype 33F (Unique to V114) | 8.3 [6.7 to 10.1] | 0.9 [0.8 to 1.0]

12. Secondary Outcome: GMFR in Serotype-specific IgG Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 and (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 1 (Shared) | 13.0 [11.0 to 15.3] | 14.4 [12.3 to 16.8]
  Serotype 3 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 3 (Shared) | 6.7 [5.8 to 7.8] | 3.9 [3.4 to 4.3]
  Serotype 4 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 4 (Shared) | 10.1 [8.6 to 11.9] | 12.4 [10.6 to 14.5]
  Serotype 5 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 5 (Shared) | 5.6 [4.8 to 6.5] | 5.2 [4.4 to 6.2]
  Serotype 6A (Shared): number analyzed (Participants) | 311 | 318
  Serotype 6A (Shared) | 30.2 [25.3 to 36.1] | 20.8 [17.5 to 24.6]
  Serotype 6B (Shared): number analyzed (Participants) | 311 | 318
  Serotype 6B (Shared) | 28.2 [23.4 to 34.1] | 17.1 [14.4 to 20.4]
  Serotype 7F (Shared): number analyzed (Participants) | 311 | 318
  Serotype 7F (Shared) | 13.6 [11.5 to 16.1] | 14.3 [12.1 to 17.0]
  Serotype 9V (Shared): number analyzed (Participants) | 311 | 318
  Serotype 9V (Shared) | 11.7 [9.9 to 13.9] | 10.3 [8.8 to 12.0]
  Serotype 14 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 14 (Shared) | 6.6 [5.4 to 7.9] | 6.3 [5.3 to 7.5]
  Serotype 18C (Shared): number analyzed (Participants) | 311 | 318
  Serotype 18C (Shared) | 22.4 [18.7 to 26.7] | 13.7 [11.6 to 16.2]
  Serotype 19A (Shared): number analyzed (Participants) | 311 | 318
  Serotype 19A (Shared) | 11.3 [9.5 to 13.5] | 9.5 [8.1 to 11.1]
  Serotype 19F (Shared): number analyzed (Participants) | 311 | 317
  Serotype 19F (Shared) | 14.2 [12.0 to 16.9] | 11.9 [10.2 to 14.0]
  Serotype 23F (Shared): number analyzed (Participants) | 311 | 318
  Serotype 23F (Shared) | 17.7 [14.7 to 21.3] | 11.0 [9.3 to 13.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 311 | 318
  Serotype 22F (Unique to V114) | 14.9 [12.4 to 18.0] | 0.9 [0.9 to 1.0]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 311 | 318
  Serotype 33F (Unique to V114) | 11.1 [9.3 to 13.1] | 0.8 [0.8 to 0.9]

13. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Titer Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using a Multiplexed Opsonophagocytic Assay. The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 307 | 314
  Serotype 1 (Shared) | 83.4 [78.7 to 87.4] | 76.1 [71.0 to 80.7]
  Serotype 3 (Shared): number analyzed (Participants) | 305 | 313
  Serotype 3 (Shared) | 72.1 [66.7 to 77.1] | 51.1 [45.4 to 56.8]
  Serotype 4 (Shared): number analyzed (Participants) | 305 | 312
  Serotype 4 (Shared) | 79.3 [74.4 to 83.7] | 84.6 [80.1 to 88.4]
  Serotype 5 (Shared): number analyzed (Participants) | 310 | 315
  Serotype 5 (Shared) | 76.8 [71.7 to 81.4] | 79.0 [74.1 to 83.4]
  Serotype 6A (Shared): number analyzed (Participants) | 279 | 283
  Serotype 6A (Shared) | 79.2 [74.0 to 83.8] | 78.1 [72.8 to 82.8]
  Serotype 6B (Shared): number analyzed (Participants) | 302 | 306
  Serotype 6B (Shared) | 83.4 [78.8 to 87.5] | 76.1 [71.0 to 80.8]
  Serotype 7F (Shared): number analyzed (Participants) | 296 | 296
  Serotype 7F (Shared) | 67.2 [61.6 to 72.5] | 65.9 [60.2 to 71.3]
  Serotype 9V (Shared): number analyzed (Participants) | 299 | 310
  Serotype 9V (Shared) | 61.2 [55.4 to 66.8] | 56.8 [51.1 to 62.4]
  Serotype 14 (Shared): number analyzed (Participants) | 304 | 308
  Serotype 14 (Shared) | 53.0 [47.2 to 58.7] | 53.2 [47.5 to 58.9]
  Serotype 18C (Shared): number analyzed (Participants) | 301 | 310
  Serotype 18C (Shared) | 83.4 [78.7 to 87.4] | 74.2 [68.9 to 79.0]
  Serotype 19A (Shared): number analyzed (Participants) | 301 | 309
  Serotype 19A (Shared) | 70.4 [64.9 to 75.5] | 69.6 [64.1 to 74.7]
  Serotype 19F (Shared): number analyzed (Participants) | 298 | 308
  Serotype 19F (Shared) | 63.4 [57.7 to 68.9] | 56.2 [50.4 to 61.8]
  Serotype 23F (Shared): number analyzed (Participants) | 284 | 288
  Serotype 23F (Shared) | 79.2 [74.0 to 83.8] | 70.8 [65.2 to 76.0]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 250 | 249
  Serotype 22F (Unique to V114) | 72.8 [66.8 to 78.2] | 16.5 [12.1 to 21.7]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 305 | 298
  Serotype 33F (Unique to V114) | 61.3 [55.6 to 66.8] | 3.0 [1.4 to 5.7]

14. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Concentration Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using an electrochemiluminescence assay. The percentage of participants who had ≥ 4-fold rise in IgG concentration are calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 1 (Shared) | 74.9 [69.7 to 79.6] | 80.8 [76.1 to 85.0]
  Serotype 3 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 3 (Shared) | 62.4 [56.7 to 67.8] | 42.8 [37.3 to 48.4]
  Serotype 4 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 4 (Shared) | 71.4 [66.0 to 76.3] | 74.2 [69.0 to 78.9]
  Serotype 5 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 5 (Shared) | 52.4 [46.7 to 58.1] | 49.4 [43.7 to 55.0]
  Serotype 6A (Shared): number analyzed (Participants) | 311 | 318
  Serotype 6A (Shared) | 88.4 [84.3 to 91.8] | 84.3 [79.8 to 88.1]
  Serotype 6B (Shared): number analyzed (Participants) | 311 | 318
  Serotype 6B (Shared) | 85.5 [81.1 to 89.2] | 77.4 [72.4 to 81.8]
  Serotype 7F (Shared): number analyzed (Participants) | 311 | 318
  Serotype 7F (Shared) | 76.8 [71.8 to 81.4] | 75.5 [70.4 to 80.1]
  Serotype 9V (Shared): number analyzed (Participants) | 311 | 318
  Serotype 9V (Shared) | 73.0 [67.7 to 77.8] | 70.4 [65.1 to 75.4]
  Serotype 14 (Shared): number analyzed (Participants) | 311 | 318
  Serotype 14 (Shared) | 54.0 [48.3 to 59.7] | 56.0 [50.3 to 61.5]
  Serotype 18C (Shared): number analyzed (Participants) | 311 | 318
  Serotype 18C (Shared) | 83.9 [79.4 to 87.8] | 75.5 [70.4 to 80.1]
  Serotype 19A (Shared): number analyzed (Participants) | 311 | 318
  Serotype 19A (Shared) | 71.4 [66.0 to 76.3] | 69.2 [63.8 to 74.2]
  Serotype 19F (Shared): number analyzed (Participants) | 311 | 317
  Serotype 19F (Shared) | 77.5 [72.4 to 82.0] | 76.3 [71.3 to 80.9]
  Serotype 23F (Shared): number analyzed (Participants) | 311 | 318
  Serotype 23F (Shared) | 79.7 [74.8 to 84.1] | 70.1 [64.8 to 75.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 311 | 318
  Serotype 22F (Unique to V114) | 76.8 [71.8 to 81.4] | 0.9 [0.2 to 2.7]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 311 | 318
  Serotype 33F (Unique to V114) | 71.1 [65.7 to 76.0] | 0.6 [0.1 to 2.3]

15. Secondary Outcome: GMT of Serotype-specific OPA at Month 12
Description: as for outcome 9
Time Frame: Month 12
Population: as for outcome 7
Measure: Number; unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 138.2 | 116.2
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 322
  Serotype 3 (Shared) | 88.3 | 56.3
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 477.2 | 666.5
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 213.4 | 209.6
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 2421.7 | 2111.3
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 2079.7 | 1453.7
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 322
  Serotype 7F (Shared) | 2161.8 | 2291.1
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 1006.8 | 1030.5
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 1543.8 | 1395.1
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 1520.4 | 1191.8
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 1724.3 | 1575.3
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 948.4 | 876.0
  Serotype 23F (Shared): number analyzed (Participants) | 320 | 323
  Serotype 23F (Shared) | 984.7 | 720.3
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 1267.4 | 99.1
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 4099.0 | 1266.6
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.19, 95% CI 2-sided [0.92 to 1.53]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.57, 95% CI 2-sided [1.29 to 1.90]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.72, 95% CI 2-sided [0.57 to 0.90]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.02, 95% CI 2-sided [0.78 to 1.33]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.15, 95% CI 2-sided [0.93 to 1.41]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.43, 95% CI 2-sided [1.16 to 1.77]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.94, 95% CI 2-sided [0.80 to 1.11]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 0.98, 95% CI 2-sided [0.81 to 1.18]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.11, 95% CI 2-sided [0.90 to 1.36]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.28, 95% CI 2-sided [1.05 to 1.55]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.09, 95% CI 2-sided [0.91 to 1.31]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.08, 95% CI 2-sided [0.91 to 1.29]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 1.37, 95% CI 2-sided [1.06 to 1.76]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 12.79, 95% CI 2-sided [9.44 to 17.34]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 3.24, 95% CI 2-sided [2.73 to 3.84]

16. Secondary Outcome: GMC of Serotype-specific IgG at Month 12
Description: as for outcome 10
Time Frame: Month 12
Population: as for outcome 7
Measure: Number; unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 1 (Shared) | 2.73 | 3.52
  Serotype 3 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 3 (Shared) | 0.39 | 0.28
  Serotype 4 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 4 (Shared) | 1.00 | 1.31
  Serotype 5 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 5 (Shared) | 2.59 | 2.91
  Serotype 6A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6A (Shared) | 4.27 | 3.13
  Serotype 6B (Shared): number analyzed (Participants) | 321 | 323
  Serotype 6B (Shared) | 5.13 | 3.46
  Serotype 7F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 7F (Shared) | 2.95 | 3.45
  Serotype 9V (Shared): number analyzed (Participants) | 321 | 323
  Serotype 9V (Shared) | 2.85 | 2.75
  Serotype 14 (Shared): number analyzed (Participants) | 321 | 323
  Serotype 14 (Shared) | 7.91 | 7.50
  Serotype 18C (Shared): number analyzed (Participants) | 321 | 323
  Serotype 18C (Shared) | 5.99 | 4.32
  Serotype 19A (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19A (Shared) | 8.19 | 7.22
  Serotype 19F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 19F (Shared) | 4.67 | 4.14
  Serotype 23F (Shared): number analyzed (Participants) | 321 | 323
  Serotype 23F (Shared) | 3.57 | 2.66
  Serotype 22F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 22F (Unique to V114) | 2.07 | 0.33
  Serotype 33F (Unique to V114): number analyzed (Participants) | 321 | 323
  Serotype 33F (Unique to V114) | 6.24 | 1.24
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.78, 95% CI 2-sided [0.65 to 0.92]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.42, 95% CI 2-sided [1.24 to 1.63]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.77, 95% CI 2-sided [0.64 to 0.91]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.89, 95% CI 2-sided [0.75 to 1.05]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.37, 95% CI 2-sided [1.12 to 1.67]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.48, 95% CI 2-sided [1.21 to 1.81]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.86, 95% CI 2-sided [0.72 to 1.02]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.04, 95% CI 2-sided [0.88 to 1.23]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.05, 95% CI 2-sided [0.88 to 1.26]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.38, 95% CI 2-sided [1.17 to 1.64]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.13, 95% CI 2-sided [0.97 to 1.33]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.13, 95% CI 2-sided [0.96 to 1.32]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.35, 95% CI 2-sided [1.12 to 1.62]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 6.20, 95% CI 2-sided [5.33 to 7.21]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 5.01, 95% CI 2-sided [4.38 to 5.73]

17. Secondary Outcome: GMFR in Serotype-specific OPA Day 1 to Month 12
Description: as for outcome 11
Time Frame: Day 1 (Baseline) and Month 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 281 | 277
  Serotype 1 (Shared) | 9.2 [7.7 to 11.1] | 7.3 [6.1 to 8.7]
  Serotype 3 (Shared): number analyzed (Participants) | 274 | 276
  Serotype 3 (Shared) | 3.0 [2.6 to 3.5] | 2.1 [1.9 to 2.4]
  Serotype 4 (Shared): number analyzed (Participants) | 276 | 277
  Serotype 4 (Shared) | 7.0 [5.8 to 8.3] | 9.4 [7.7 to 11.3]
  Serotype 5 (Shared): number analyzed (Participants) | 281 | 280
  Serotype 5 (Shared) | 5.5 [4.6 to 6.7] | 5.7 [4.7 to 6.9]
  Serotype 6A (Shared): number analyzed (Participants) | 255 | 254
  Serotype 6A (Shared) | 5.7 [4.9 to 6.8] | 4.9 [4.2 to 5.7]
  Serotype 6B (Shared): number analyzed (Participants) | 272 | 273
  Serotype 6B (Shared) | 10.4 [8.4 to 12.7] | 7.3 [6.1 to 8.8]
  Serotype 7F (Shared): number analyzed (Participants) | 270 | 262
  Serotype 7F (Shared) | 4.6 [3.8 to 5.5] | 4.9 [4.1 to 6.0]
  Serotype 9V (Shared): number analyzed (Participants) | 272 | 275
  Serotype 9V (Shared) | 2.7 [2.3 to 3.1] | 2.7 [2.3 to 3.1]
  Serotype 14 (Shared): number analyzed (Participants) | 274 | 270
  Serotype 14 (Shared) | 3.9 [3.3 to 4.7] | 3.5 [2.9 to 4.2]
  Serotype 18C (Shared): number analyzed (Participants) | 275 | 274
  Serotype 18C (Shared) | 6.5 [5.6 to 7.6] | 5.2 [4.5 to 6.1]
  Serotype 19A (Shared): number analyzed (Participants) | 269 | 276
  Serotype 19A (Shared) | 4.9 [4.1 to 5.9] | 4.3 [3.6 to 5.0]
  Serotype 19F (Shared): number analyzed (Participants) | 267 | 272
  Serotype 19F (Shared) | 3.0 [2.6 to 3.5] | 2.8 [2.5 to 3.3]
  Serotype 23F (Shared): number analyzed (Participants) | 255 | 256
  Serotype 23F (Shared) | 7.1 [5.8 to 8.7] | 5.1 [4.2 to 6.3]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 225 | 213
  Serotype 22F (Unique to V114) | 12.3 [9.3 to 16.3] | 1.3 [1.0 to 1.6]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 278 | 269
  Serotype 33F (Unique to V114) | 3.0 [2.5 to 3.6] | 0.9 [0.8 to 1.0]

18. Secondary Outcome: GMFR in Serotype-specific IgG Day 1 to Month 12
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Month 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 1 (Shared) | 5.2 [4.5 to 6.0] | 6.6 [5.7 to 7.7]
  Serotype 3 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 3 (Shared) | 2.6 [2.3 to 2.9] | 1.8 [1.7 to 2.0]
  Serotype 4 (Shared): number analyzed (Participants) | 282 | 281
  Serotype 4 (Shared) | 4.3 [3.8 to 4.9] | 5.5 [4.8 to 6.3]
  Serotype 5 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 5 (Shared) | 2.7 [2.4 to 3.0] | 3.0 [2.6 to 3.4]
  Serotype 6A (Shared): number analyzed (Participants) | 282 | 282
  Serotype 6A (Shared) | 11.1 [9.5 to 13.0] | 8.1 [6.9 to 9.3]
  Serotype 6B (Shared): number analyzed (Participants) | 282 | 282
  Serotype 6B (Shared) | 10.3 [8.7 to 12.2] | 7.2 [6.2 to 8.4]
  Serotype 7F (Shared): number analyzed (Participants) | 282 | 282
  Serotype 7F (Shared) | 5.5 [4.8 to 6.2] | 6.4 [5.5 to 7.5]
  Serotype 9V (Shared): number analyzed (Participants) | 282 | 282
  Serotype 9V (Shared) | 5.6 [4.9 to 6.4] | 5.4 [4.7 to 6.1]
  Serotype 14 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 14 (Shared) | 3.9 [3.4 to 4.6] | 4.1 [3.5 to 4.7]
  Serotype 18C (Shared): number analyzed (Participants) | 282 | 282
  Serotype 18C (Shared) | 8.0 [6.9 to 9.3] | 5.6 [4.9 to 6.5]
  Serotype 19A (Shared): number analyzed (Participants) | 282 | 282
  Serotype 19A (Shared) | 4.9 [4.3 to 5.6] | 4.3 [3.8 to 4.9]
  Serotype 19F (Shared): number analyzed (Participants) | 281 | 281
  Serotype 19F (Shared) | 5.2 [4.6 to 6.0] | 4.9 [4.3 to 5.6]
  Serotype 23F (Shared): number analyzed (Participants) | 282 | 282
  Serotype 23F (Shared) | 6.6 [5.7 to 7.6] | 4.9 [4.3 to 5.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 282 | 282
  Serotype 22F (Unique to V114) | 6.0 [5.1 to 7.0] | 1.0 [0.9 to 1.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 282 | 282
  Serotype 33F (Unique to V114) | 4.7 [4.1 to 5.4] | 0.9 [0.9 to 1.0]

19. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Titer Day 1 to Month 12
Description: as for outcome 13
Time Frame: Day 1 (Baseline) and Month 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 281 | 277
  Serotype 1 (Shared) | 69.4 [63.6 to 74.7] | 61.4 [55.4 to 67.1]
  Serotype 3 (Shared): number analyzed (Participants) | 274 | 276
  Serotype 3 (Shared) | 39.4 [33.6 to 45.5] | 25.7 [20.7 to 31.3]
  Serotype 4 (Shared): number analyzed (Participants) | 276 | 277
  Serotype 4 (Shared) | 63.0 [57.1 to 68.8] | 67.1 [61.3 to 72.6]
  Serotype 5 (Shared): number analyzed (Participants) | 281 | 280
  Serotype 5 (Shared) | 58.4 [52.4 to 64.2] | 57.5 [51.5 to 63.4]
  Serotype 6A (Shared): number analyzed (Participants) | 255 | 254
  Serotype 6A (Shared) | 61.2 [54.9 to 67.2] | 54.3 [48.0 to 60.6]
  Serotype 6B (Shared): number analyzed (Participants) | 272 | 273
  Serotype 6B (Shared) | 68.8 [62.9 to 74.2] | 60.4 [54.4 to 66.3]
  Serotype 7F (Shared): number analyzed (Participants) | 270 | 262
  Serotype 7F (Shared) | 50.4 [44.2 to 56.5] | 48.9 [42.7 to 55.1]
  Serotype 9V (Shared): number analyzed (Participants) | 272 | 275
  Serotype 9V (Shared) | 34.6 [28.9 to 40.5] | 32.0 [26.5 to 37.9]
  Serotype 14 (Shared): number analyzed (Participants) | 274 | 270
  Serotype 14 (Shared) | 41.6 [35.7 to 47.7] | 42.2 [36.3 to 48.4]
  Serotype 18C (Shared): number analyzed (Participants) | 275 | 274
  Serotype 18C (Shared) | 63.3 [57.3 to 69.0] | 54.4 [48.3 to 60.4]
  Serotype 19A (Shared): number analyzed (Participants) | 269 | 276
  Serotype 19A (Shared) | 53.2 [47.0 to 59.2] | 47.5 [41.4 to 53.5]
  Serotype 19F (Shared): number analyzed (Participants) | 267 | 272
  Serotype 19F (Shared) | 41.2 [35.2 to 47.4] | 35.3 [29.6 to 41.3]
  Serotype 23F (Shared): number analyzed (Participants) | 255 | 256
  Serotype 23F (Shared) | 62.4 [56.1 to 68.3] | 53.5 [47.2 to 59.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 225 | 213
  Serotype 22F (Unique to V114) | 64.0 [57.4 to 70.3] | 14.1 [9.7 to 19.5]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 278 | 269
  Serotype 33F (Unique to V114) | 34.5 [29.0 to 40.4] | 4.8 [2.6 to 8.1]

20. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Concentration Day 1 to Month 12
Description: as for outcome 14
Time Frame: Day 1 (Baseline) and Month 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 1 (Shared) | 56.0 [50.0 to 61.9] | 65.6 [59.7 to 71.1]
  Serotype 3 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 3 (Shared) | 27.0 [21.9 to 32.5] | 12.4 [8.8 to 16.8]
  Serotype 4 (Shared): number analyzed (Participants) | 282 | 281
  Serotype 4 (Shared) | 47.2 [41.2 to 53.2] | 57.7 [51.6 to 63.5]
  Serotype 5 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 5 (Shared) | 30.9 [25.5 to 36.6] | 34.4 [28.9 to 40.3]
  Serotype 6A (Shared): number analyzed (Participants) | 282 | 282
  Serotype 6A (Shared) | 75.5 [70.1 to 80.4] | 66.7 [60.8 to 72.1]
  Serotype 6B (Shared): number analyzed (Participants) | 282 | 282
  Serotype 6B (Shared) | 73.0 [67.5 to 78.1] | 62.1 [56.1 to 67.7]
  Serotype 7F (Shared): number analyzed (Participants) | 282 | 282
  Serotype 7F (Shared) | 59.9 [54.0 to 65.7] | 64.9 [59.0 to 70.5]
  Serotype 9V (Shared): number analyzed (Participants) | 282 | 282
  Serotype 9V (Shared) | 60.6 [54.7 to 66.4] | 55.3 [49.3 to 61.2]
  Serotype 14 (Shared): number analyzed (Participants) | 282 | 282
  Serotype 14 (Shared) | 42.6 [36.7 to 48.6] | 46.8 [40.9 to 52.8]
  Serotype 18C (Shared): number analyzed (Participants) | 282 | 282
  Serotype 18C (Shared) | 70.2 [64.5 to 75.5] | 58.5 [52.5 to 64.3]
  Serotype 19A (Shared): number analyzed (Participants) | 282 | 282
  Serotype 19A (Shared) | 53.9 [47.9 to 59.8] | 50.0 [44.0 to 56.0]
  Serotype 19F (Shared): number analyzed (Participants) | 281 | 281
  Serotype 19F (Shared) | 56.9 [50.9 to 62.8] | 52.3 [46.3 to 58.3]
  Serotype 23F (Shared): number analyzed (Participants) | 282 | 282
  Serotype 23F (Shared) | 59.6 [53.6 to 65.4] | 51.4 [45.4 to 57.4]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 282 | 282
  Serotype 22F (Unique to V114) | 58.9 [52.9 to 64.7] | 1.8 [0.6 to 4.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 282 | 282
  Serotype 33F (Unique to V114) | 52.5 [46.5 to 58.4] | 1.1 [0.2 to 3.1]

21. Secondary Outcome: GMFR in Serotype-specific OPA Day 1 to Month 13
Description: as for outcome 11
Time Frame: Day 1 (Baseline) and Month 13
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 272 | 269
  Serotype 1 (Shared) | 24.7 [20.7 to 29.4] | 15.5 [12.9 to 18.5]
  Serotype 3 (Shared): number analyzed (Participants) | 268 | 267
  Serotype 3 (Shared) | 9.1 [7.9 to 10.5] | 8.7 [7.5 to 10.0]
  Serotype 4 (Shared): number analyzed (Participants) | 270 | 268
  Serotype 4 (Shared) | 23.8 [19.5 to 29.2] | 21.5 [17.5 to 26.3]
  Serotype 5 (Shared): number analyzed (Participants) | 273 | 272
  Serotype 5 (Shared) | 17.2 [14.1 to 21.1] | 14.5 [12.0 to 17.5]
  Serotype 6A (Shared): number analyzed (Participants) | 243 | 245
  Serotype 6A (Shared) | 7.7 [6.5 to 9.2] | 6.3 [5.4 to 7.3]
  Serotype 6B (Shared): number analyzed (Participants) | 264 | 266
  Serotype 6B (Shared) | 16.2 [13.3 to 19.8] | 14.3 [11.7 to 17.4]
  Serotype 7F (Shared): number analyzed (Participants) | 262 | 254
  Serotype 7F (Shared) | 11.0 [9.0 to 13.4] | 10.2 [8.2 to 12.5]
  Serotype 9V (Shared): number analyzed (Participants) | 265 | 266
  Serotype 9V (Shared) | 5.2 [4.5 to 6.1] | 4.6 [3.9 to 5.3]
  Serotype 14 (Shared): number analyzed (Participants) | 268 | 264
  Serotype 14 (Shared) | 8.2 [6.8 to 9.8] | 6.7 [5.6 to 8.0]
  Serotype 18C (Shared): number analyzed (Participants) | 267 | 266
  Serotype 18C (Shared) | 10.1 [8.6 to 11.7] | 9.0 [7.7 to 10.4]
  Serotype 19A (Shared): number analyzed (Participants) | 262 | 267
  Serotype 19A (Shared) | 10.4 [8.5 to 12.6] | 8.5 [7.2 to 10.2]
  Serotype 19F (Shared): number analyzed (Participants) | 263 | 264
  Serotype 19F (Shared) | 7.0 [6.0 to 8.1] | 6.3 [5.5 to 7.2]
  Serotype 23F (Shared): number analyzed (Participants) | 250 | 249
  Serotype 23F (Shared) | 12.6 [10.3 to 15.5] | 9.7 [7.8 to 12.0]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 224 | 230
  Serotype 22F (Unique to V114) | 30.2 [22.7 to 40.1] | 16.2 [11.8 to 22.2]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 269 | 258
  Serotype 33F (Unique to V114) | 5.8 [4.8 to 7.0] | 5.5 [4.5 to 6.7]

22. Secondary Outcome: GMFR in Serotype-specific IgG Day 1 to Month 13
Description: as for outcome 18
Time Frame: Day 1 (Baseline) and Month 13
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 1 (Shared) | 9.9 [8.7 to 11.4] | 10.5 [9.1 to 12.2]
  Serotype 3 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 3 (Shared) | 6.9 [6.0 to 7.8] | 6.7 [6.0 to 7.6]
  Serotype 4 (Shared): number analyzed (Participants) | 273 | 273
  Serotype 4 (Shared) | 8.6 [7.6 to 9.8] | 9.5 [8.3 to 11.0]
  Serotype 5 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 5 (Shared) | 5.9 [5.2 to 6.8] | 5.9 [5.2 to 6.8]
  Serotype 6A (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6A (Shared) | 13.1 [11.2 to 15.3] | 10.8 [9.3 to 12.5]
  Serotype 6B (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6B (Shared) | 13.7 [11.7 to 16.1] | 11.9 [10.2 to 13.9]
  Serotype 7F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 7F (Shared) | 11.1 [9.8 to 12.7] | 11.2 [9.7 to 12.9]
  Serotype 9V (Shared): number analyzed (Participants) | 273 | 274
  Serotype 9V (Shared) | 9.8 [8.5 to 11.3] | 9.2 [8.0 to 10.5]
  Serotype 14 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 14 (Shared) | 7.4 [6.3 to 8.7] | 6.9 [5.9 to 8.1]
  Serotype 18C (Shared): number analyzed (Participants) | 273 | 274
  Serotype 18C (Shared) | 9.8 [8.5 to 11.3] | 8.2 [7.1 to 9.4]
  Serotype 19A (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19A (Shared) | 7.9 [6.9 to 9.0] | 7.0 [6.1 to 8.0]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 273
  Serotype 19F (Shared) | 10.7 [9.3 to 12.4] | 10.0 [8.6 to 11.5]
  Serotype 23F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 23F (Shared) | 9.1 [7.9 to 10.5] | 7.6 [6.6 to 8.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 273 | 274
  Serotype 22F (Unique to V114) | 14.2 [12.0 to 16.7] | 10.0 [8.4 to 12.0]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 273 | 274
  Serotype 33F (Unique to V114) | 8.1 [7.1 to 9.2] | 10.1 [8.6 to 11.8]

23. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Titer Day 1 to Month 13
Description: as for outcome 13
Time Frame: Day 1 (Baseline) and Month 13
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 272 | 269
  Serotype 1 (Shared) | 87.9 [83.4 to 91.5] | 78.8 [73.4 to 83.5]
  Serotype 3 (Shared): number analyzed (Participants) | 268 | 267
  Serotype 3 (Shared) | 78.7 [73.3 to 83.5] | 76.0 [70.4 to 81.0]
  Serotype 4 (Shared): number analyzed (Participants) | 270 | 268
  Serotype 4 (Shared) | 83.7 [78.7 to 87.9] | 84.3 [79.4 to 88.5]
  Serotype 5 (Shared): number analyzed (Participants) | 273 | 272
  Serotype 5 (Shared) | 79.9 [74.6 to 84.4] | 80.9 [75.7 to 85.4]
  Serotype 6A (Shared): number analyzed (Participants) | 243 | 245
  Serotype 6A (Shared) | 68.3 [62.1 to 74.1] | 64.5 [58.1 to 70.5]
  Serotype 6B (Shared): number analyzed (Participants) | 264 | 266
  Serotype 6B (Shared) | 78.0 [72.5 to 82.9] | 77.1 [71.5 to 82.0]
  Serotype 7F (Shared): number analyzed (Participants) | 262 | 254
  Serotype 7F (Shared) | 72.1 [66.3 to 77.5] | 64.6 [58.3 to 70.4]
  Serotype 9V (Shared): number analyzed (Participants) | 265 | 266
  Serotype 9V (Shared) | 55.8 [49.6 to 61.9] | 50.8 [44.6 to 56.9]
  Serotype 14 (Shared): number analyzed (Participants) | 268 | 264
  Serotype 14 (Shared) | 63.8 [57.7 to 69.6] | 58.7 [52.5 to 64.7]
  Serotype 18C (Shared): number analyzed (Participants) | 267 | 266
  Serotype 18C (Shared) | 75.7 [70.1 to 80.7] | 73.7 [68.0 to 78.9]
  Serotype 19A (Shared): number analyzed (Participants) | 262 | 267
  Serotype 19A (Shared) | 70.2 [64.3 to 75.7] | 66.3 [60.3 to 71.9]
  Serotype 19F (Shared): number analyzed (Participants) | 263 | 264
  Serotype 19F (Shared) | 68.4 [62.4 to 74.0] | 62.1 [56.0 to 68.0]
  Serotype 23F (Shared): number analyzed (Participants) | 250 | 249
  Serotype 23F (Shared) | 74.4 [68.5 to 79.7] | 66.3 [60.0 to 72.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 224 | 230
  Serotype 22F (Unique to V114) | 79.5 [73.6 to 84.6] | 62.6 [56.0 to 68.9]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 269 | 258
  Serotype 33F (Unique to V114) | 55.8 [49.6 to 61.8] | 51.6 [45.3 to 57.8]

24. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Concentration Day 1 to Month 13
Description: as for outcome 14
Time Frame: Day 1 (Baseline) and Month 13
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 1 (Shared) | 79.5 [74.2 to 84.1] | 78.5 [73.1 to 83.2]
  Serotype 3 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 3 (Shared) | 72.5 [66.8 to 77.7] | 68.6 [62.8 to 74.1]
  Serotype 4 (Shared): number analyzed (Participants) | 273 | 273
  Serotype 4 (Shared) | 76.6 [71.1 to 81.5] | 75.5 [69.9 to 80.4]
  Serotype 5 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 5 (Shared) | 59.7 [53.6 to 65.6] | 59.9 [53.8 to 65.7]
  Serotype 6A (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6A (Shared) | 81.0 [75.8 to 85.4] | 77.0 [71.6 to 81.9]
  Serotype 6B (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6B (Shared) | 81.0 [75.8 to 85.4] | 77.0 [71.6 to 81.9]
  Serotype 7F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 7F (Shared) | 81.7 [76.6 to 86.1] | 81.4 [76.3 to 85.8]
  Serotype 9V (Shared): number analyzed (Participants) | 273 | 274
  Serotype 9V (Shared) | 76.2 [70.7 to 81.1] | 73.4 [67.7 to 78.5]
  Serotype 14 (Shared): number analyzed (Participants) | 273 | 274
  Serotype 14 (Shared) | 68.5 [62.6 to 74.0] | 63.9 [57.9 to 69.6]
  Serotype 18C (Shared): number analyzed (Participants) | 273 | 274
  Serotype 18C (Shared) | 78.0 [72.6 to 82.8] | 70.8 [65.0 to 76.1]
  Serotype 19A (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19A (Shared) | 70.0 [64.1 to 75.3] | 66.4 [60.5 to 72.0]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 273
  Serotype 19F (Shared) | 77.3 [71.9 to 82.1] | 74.0 [68.4 to 79.1]
  Serotype 23F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 23F (Shared) | 72.2 [66.4 to 77.4] | 69.7 [63.9 to 75.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 273 | 274
  Serotype 22F (Unique to V114) | 80.6 [75.4 to 85.1] | 71.9 [66.2 to 77.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 273 | 274
  Serotype 33F (Unique to V114) | 75.5 [69.9 to 80.4] | 76.6 [71.2 to 81.5]

25. Secondary Outcome: GMFR in Serotype-specific OPA Month 12 to Month 13
Description: as for outcome 11
Time Frame: Month 12 (Baseline) and Month 13
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 273 | 270
  Serotype 1 (Shared) | 2.7 [2.4 to 3.0] | 2.3 [2.0 to 2.6]
  Serotype 3 (Shared): number analyzed (Participants) | 267 | 270
  Serotype 3 (Shared) | 3.0 [2.7 to 3.4] | 4.1 [3.6 to 4.6]
  Serotype 4 (Shared): number analyzed (Participants) | 273 | 273
  Serotype 4 (Shared) | 3.3 [2.9 to 3.9] | 2.3 [2.0 to 2.6]
  Serotype 5 (Shared): number analyzed (Participants) | 275 | 274
  Serotype 5 (Shared) | 3.1 [2.7 to 3.5] | 2.6 [2.3 to 2.9]
  Serotype 6A (Shared): number analyzed (Participants) | 264 | 268
  Serotype 6A (Shared) | 1.3 [1.2 to 1.5] | 1.3 [1.2 to 1.5]
  Serotype 6B (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6B (Shared) | 1.5 [1.4 to 1.7] | 1.9 [1.8 to 2.2]
  Serotype 7F (Shared): number analyzed (Participants) | 275 | 274
  Serotype 7F (Shared) | 2.3 [2.1 to 2.6] | 2.1 [1.9 to 2.3]
  Serotype 9V (Shared): number analyzed (Participants) | 274 | 273
  Serotype 9V (Shared) | 2.0 [1.8 to 2.2] | 1.7 [1.6 to 2.0]
  Serotype 14 (Shared): number analyzed (Participants) | 272 | 272
  Serotype 14 (Shared) | 2.1 [1.9 to 2.4] | 1.9 [1.7 to 2.1]
  Serotype 18C (Shared): number analyzed (Participants) | 272 | 274
  Serotype 18C (Shared) | 1.5 [1.4 to 1.7] | 1.7 [1.5 to 1.9]
  Serotype 19A (Shared): number analyzed (Participants) | 270 | 273
  Serotype 19A (Shared) | 2.1 [1.9 to 2.4] | 2.0 [1.8 to 2.3]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19F (Shared) | 2.3 [2.0 to 2.6] | 2.3 [2.1 to 2.6]
  Serotype 23F (Shared): number analyzed (Participants) | 268 | 270
  Serotype 23F (Shared) | 1.9 [1.6 to 2.1] | 1.9 [1.7 to 2.2]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 265 | 245
  Serotype 22F (Unique to V114) | 2.5 [2.1 to 2.9] | 14.2 [10.6 to 19.0]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 271 | 263
  Serotype 33F (Unique to V114) | 2.0 [1.8 to 2.2] | 6.2 [5.2 to 7.5]

26. Secondary Outcome: GMFR in Serotype-specific IgG Month 12 to Month 13
Description: as for outcome 18
Time Frame: Month 12 (Baseline) and Month 13
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 1 (Shared) | 1.9 [1.8 to 2.1] | 1.6 [1.5 to 1.7]
  Serotype 3 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 3 (Shared) | 2.6 [2.4 to 2.9] | 3.7 [3.3 to 4.1]
  Serotype 4 (Shared): number analyzed (Participants) | 274 | 272
  Serotype 4 (Shared) | 2.0 [1.8 to 2.2] | 1.7 [1.6 to 1.9]
  Serotype 5 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 5 (Shared) | 2.3 [2.1 to 2.5] | 2.0 [1.8 to 2.1]
  Serotype 6A (Shared): number analyzed (Participants) | 274 | 274
  Serotype 6A (Shared) | 1.2 [1.1 to 1.2] | 1.3 [1.3 to 1.4]
  Serotype 6B (Shared): number analyzed (Participants) | 274 | 274
  Serotype 6B (Shared) | 1.3 [1.2 to 1.4] | 1.6 [1.5 to 1.8]
  Serotype 7F (Shared): number analyzed (Participants) | 274 | 274
  Serotype 7F (Shared) | 2.1 [1.9 to 2.2] | 1.8 [1.6 to 1.9]
  Serotype 9V (Shared): number analyzed (Participants) | 274 | 274
  Serotype 9V (Shared) | 1.8 [1.6 to 1.9] | 1.7 [1.6 to 1.9]
  Serotype 14 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 14 (Shared) | 1.9 [1.7 to 2.1] | 1.7 [1.6 to 1.8]
  Serotype 18C (Shared): number analyzed (Participants) | 274 | 274
  Serotype 18C (Shared) | 1.2 [1.2 to 1.3] | 1.5 [1.4 to 1.6]
  Serotype 19A (Shared): number analyzed (Participants) | 274 | 274
  Serotype 19A (Shared) | 1.6 [1.5 to 1.7] | 1.6 [1.5 to 1.7]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19F (Shared) | 2.0 [1.9 to 2.2] | 2.1 [1.9 to 2.3]
  Serotype 23F (Shared): number analyzed (Participants) | 274 | 274
  Serotype 23F (Shared) | 1.4 [1.3 to 1.5] | 1.6 [1.5 to 1.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 274 | 274
  Serotype 22F (Unique to V114) | 2.4 [2.2 to 2.6] | 10.0 [8.4 to 11.9]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 274 | 274
  Serotype 33F (Unique to V114) | 1.7 [1.6 to 1.9] | 10.7 [9.1 to 12.5]

27. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Titer Month 12 to Month 13
Description: as for outcome 13
Time Frame: Month 12 (Baseline) and Month 13
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 273 | 270
  Serotype 1 (Shared) | 29.7 [24.3 to 35.5] | 25.6 [20.5 to 31.2]
  Serotype 3 (Shared): number analyzed (Participants) | 267 | 270
  Serotype 3 (Shared) | 39.0 [33.1 to 45.1] | 49.6 [43.5 to 55.8]
  Serotype 4 (Shared): number analyzed (Participants) | 273 | 273
  Serotype 4 (Shared) | 36.3 [30.6 to 42.3] | 22.3 [17.5 to 27.8]
  Serotype 5 (Shared): number analyzed (Participants) | 275 | 274
  Serotype 5 (Shared) | 34.9 [29.3 to 40.9] | 29.2 [23.9 to 35.0]
  Serotype 6A (Shared): number analyzed (Participants) | 264 | 268
  Serotype 6A (Shared) | 9.1 [5.9 to 13.2] | 10.4 [7.1 to 14.7]
  Serotype 6B (Shared): number analyzed (Participants) | 273 | 274
  Serotype 6B (Shared) | 8.8 [5.7 to 12.8] | 16.1 [11.9 to 21.0]
  Serotype 7F (Shared): number analyzed (Participants) | 275 | 274
  Serotype 7F (Shared) | 24.7 [19.7 to 30.3] | 21.2 [16.5 to 26.5]
  Serotype 9V (Shared): number analyzed (Participants) | 274 | 273
  Serotype 9V (Shared) | 20.1 [15.5 to 25.3] | 16.5 [12.3 to 21.4]
  Serotype 14 (Shared): number analyzed (Participants) | 272 | 272
  Serotype 14 (Shared) | 21.3 [16.6 to 26.7] | 12.9 [9.1 to 17.4]
  Serotype 18C (Shared): number analyzed (Participants) | 272 | 274
  Serotype 18C (Shared) | 10.7 [7.3 to 15.0] | 15.7 [11.6 to 20.6]
  Serotype 19A (Shared): number analyzed (Participants) | 270 | 273
  Serotype 19A (Shared) | 20.4 [15.7 to 25.7] | 17.9 [13.6 to 23.0]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19F (Shared) | 25.3 [20.2 to 30.9] | 27.4 [22.2 to 33.1]
  Serotype 23F (Shared): number analyzed (Participants) | 268 | 270
  Serotype 23F (Shared) | 19.0 [14.5 to 24.2] | 17.8 [13.4 to 22.9]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 265 | 245
  Serotype 22F (Unique to V114) | 26.8 [21.6 to 32.6] | 62.0 [55.6 to 68.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 271 | 263
  Serotype 33F (Unique to V114) | 22.1 [17.3 to 27.6] | 54.4 [48.1 to 60.5]

28. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Concentration Month 12 to Month 13
Description: as for outcome 14
Time Frame: Month 12 (Baseline) and Month 13
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 326 | 325
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 1 (Shared) | 15.0 [11.0 to 19.7] | 8.8 [5.7 to 12.8]
  Serotype 3 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 3 (Shared) | 31.4 [25.9 to 37.2] | 43.8 [37.8 to 49.9]
  Serotype 4 (Shared): number analyzed (Participants) | 274 | 272
  Serotype 4 (Shared) | 14.2 [10.3 to 18.9] | 8.8 [5.7 to 12.8]
  Serotype 5 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 5 (Shared) | 20.1 [15.5 to 25.3] | 15.0 [11.0 to 19.7]
  Serotype 6A (Shared): number analyzed (Participants) | 274 | 274
  Serotype 6A (Shared) | 1.1 [0.2 to 3.2] | 4.4 [2.3 to 7.5]
  Serotype 6B (Shared): number analyzed (Participants) | 274 | 274
  Serotype 6B (Shared) | 4.7 [2.6 to 8.0] | 11.3 [7.8 to 15.7]
  Serotype 7F (Shared): number analyzed (Participants) | 274 | 274
  Serotype 7F (Shared) | 17.2 [12.9 to 22.1] | 10.2 [6.9 to 14.4]
  Serotype 9V (Shared): number analyzed (Participants) | 274 | 274
  Serotype 9V (Shared) | 10.6 [7.2 to 14.8] | 9.1 [6.0 to 13.2]
  Serotype 14 (Shared): number analyzed (Participants) | 274 | 274
  Serotype 14 (Shared) | 14.2 [10.3 to 18.9] | 9.5 [6.3 to 13.6]
  Serotype 18C (Shared): number analyzed (Participants) | 274 | 274
  Serotype 18C (Shared) | 0.4 [0.0 to 2.0] | 6.9 [4.2 to 10.6]
  Serotype 19A (Shared): number analyzed (Participants) | 274 | 274
  Serotype 19A (Shared) | 8.0 [5.1 to 11.9] | 7.7 [4.8 to 11.5]
  Serotype 19F (Shared): number analyzed (Participants) | 273 | 274
  Serotype 19F (Shared) | 13.9 [10.0 to 18.6] | 17.9 [13.5 to 22.9]
  Serotype 22F (Shared): number analyzed (Participants) | 274 | 274
  Serotype 22F (Shared) | 3.6 [1.8 to 6.6] | 10.2 [6.9 to 14.4]
  Serotype 23F (Unique to V114): number analyzed (Participants) | 274 | 274
  Serotype 23F (Unique to V114) | 21.5 [16.8 to 26.9] | 71.2 [65.4 to 76.5]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 274 | 274
  Serotype 33F (Unique to V114) | 10.6 [7.2 to 14.8] | 77.0 [71.6 to 81.9]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after each vaccination; Serious adverse events and all-cause mortality: Up to Month 13 (Up to 44 days after vaccination 2)
Description: The analysis population included all randomized participants who received study intervention at the specified timepoint. Adverse events were reported (1) following administration of either V114 or Prevnar 13™ and (2) following administration of PNEUMOVAX™23.
Groups:
- V114 (Post-PNEUMOVAX™23): Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
- Prevnar 13™ (Post-PNEUMOVAX™23): Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 12 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™ | V114 (Post-PNEUMOVAX™23) | Prevnar 13™ (Post-PNEUMOVAX™23)
All-Cause Mortality (participants affected / at risk) | 0/327 | 0/324 | 0/298 | 0/302
Serious Adverse Events (participants affected / at risk) | 17/327 | 19/324 | 1/298 | 2/302
Other Adverse Events (participants affected / at risk) | 221/327 | 181/324 | 217/298 | 210/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=327) | Prevnar 13™ (N=324) | V114 (Post-PNEUMOVAX™23) (N=298) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=302)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hangover (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=327) | Prevnar 13™ (N=324) | V114 (Post-PNEUMOVAX™23) (N=298) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=302)
Fatigue (General disorders) | 77 (89) | 45 (53) | 77 (103) | 66 (77)
Injection site erythema (General disorders) | 39 (41) | 26 (28) | 53 (57) | 51 (53)
Injection site pain (General disorders) | 181 (204) | 137 (155) | 186 (210) | 177 (210)
Injection site swelling (General disorders) | 54 (55) | 40 (43) | 84 (85) | 79 (82)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (26) | 17 (19) | 25 (34) | 25 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 58 (62) | 36 (39) | 64 (71) | 50 (55)
Headache (Nervous system disorders) | 46 (58) | 41 (52) | 36 (43) | 38 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03480763/Prot_SAP_000.pdf